CLINICAL TRIAL: NCT03831490
Title: IMPACT - Study for Improving Maternal, Pregnancy and Child Outcomes
Brief Title: Study for Improving Maternal, Pregnancy and Child Outcomes
Acronym: IMPACT
Status: Completed | Type: Observational
Sponsor: Uppsala University (Other)
Collaborators: Thermo Fisher Scientific, Inc (Industry); Perkin Elmer Inc. (Industry); Roche Pharma AG (Industry)
Responsible Party: Sponsor
Other Study IDs: Dnr 2018-231
Record Dates: First submitted 2019-02-01; First posted 2019-02-05 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Pre-Eclampsia
Keywords: screening; biomarkers; prediction
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 9 Months
Biospecimen Retention: Samples With DNA — At centers with biobank possibilities, serum, plasma and buffy-coat samples will be collected at the same time as the serum sample for analyze of Placental Growth Factor. The samples for the biobank will be stored for future research related to prediction, diagnosis and prevention of pregnancy complications.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: history — combining these 4 interventions will great an algorithm predicting preeclampsia
  Other Names: mean material blod pressure; PlGF - blood sample; a- uterine doppler

SUMMARY:
The overall aims of this proposal are to improve, facilitate, optimize and equalize the existing screening system for adverse pregnancy outcomes in early pregnancy in order to limit adverse consequences for both the mother and infant, by:

1. Creating a Swedish prediction model with population-specific risk factors, optimized for the Swedish health care system, identifying high-risk women for preterm preeclampsia and validate the model within the cohort. This would give us the possibility to start aspirin prophylaxis in time, which has been proven to reduce the risk of developing preterm preeclampsia by 50%.
2. Validating the Fetal Medicine Foundation prediction model for detection of preterm (< 37 gestational weeks) preeclampsia in a Swedish population.
3. Creating a prediction model identifying high-risk women for overall preeclampsia during pregnancy and birth of a small for gestational age infant in order to plan individualized surveillance for early detection, which has been proven beneficial for both the mother and infant.
4. Creating a national pregnancy biobank with blood samples and individual clinical registry data, including pregnancy outcomes, enabling future research on prevention and early detection for various adverse pregnancy outcomes which could be such as preterm birth and intrauterine growth restriction.

DETAILED DESCRIPTION:
Preeclampsia is a pregnancy-specific syndrome that affects 3-5% of all pregnancies and traditionally defined as new onset hypertension (blood pressure ≥ 140/90) and proteinuria after gestational week 20. The syndrome is one of the leading causes of maternal and perinatal acute morbidity and long-term disability and accounts for about 50 000 maternal deaths annually worldwide. Morbidity risks for the mother include seizures, intracranial hemorrhage, kidney failure, heart failure and pulmonary edema. Risks for the fetus include fetal growth restriction, preterm birth and hypoxia. Generally preterm preeclampsia (delivery before 37 weeks) is more severe than term preeclampsia.

Risk assessment for preeclampsia enables both prevention and early prediction of the disease.

Swedish risk assessment for preeclampsia in early pregnancy is still obtained by maternal history and characteristics, without medical examinations, which only detects about 30% of women that will develop preeclampsia. Risk factors are evaluated individually without being incorporated into a combined model that would allow multivariable analysis. This approach has been proven to be poor due to low specificity and sensitivity. Lately a more complex prediction model has been developed by the Fetal Medicine Foundation, using multivariable analysis and including serum biomarkers and physiological measurements reflecting maternal adaption to pregnancy. Intervention with aspirin given to identified high-risk pregnancies according this model has been shown to decrease the incidence of preterm (< 37 gestational weeks) preeclampsia (OR: 0.38; 95% CI 0.20-0.74), compared to placebo. Detection rates and cut-off values have been shown to vary between populations, depending on differences in population characteristics and incidence of disease, overfitting of the original model and differences in healthcare systems. Therefore, the model needs to be validated in Sweden. Further, the Fetal Medicine Foundation prediction model includes expensive covariates such as several biochemical markers and uterine artery Doppler. There is a need to create, validate and implement a cost-effective prediction model for first trimester screening for preeclampsia in a Swedish population, with the purpose to select who might benefit from aspirin prophylaxis to prevent preterm preeclampsia. We will study preeclampsia both according to the definition used in Sweden prior to 2020 and the definition used hereafter.

Early detection of preeclampsia remains one of the major focuses of maternal health care and is emphasized by the WHO, since it has proven to be beneficial for both the mother and unborn child. Small-for-gestational-age fetuses not identified before delivery have an increased risk of adverse perinatal outcomes, compared to those identified during pregnancy. Identification of high-risk pregnancies is therefore important in early pregnancy not only to plan for prophylactic interventions, but also to optimize surveillance and to plan deliveries. Today most Swedish women attend the same maternal health care program with increasing number of visits in the end of pregnancy. By risk identification in early pregnancy we can individualize maternal health care and target women at high risk early in pregnancy. High-risk pregnancies can be referred to specialized health care and normal pregnancies followed at the basic maternal health care.

The Swedish registry data is unique and combining it with a biobank containing blood samples from the first trimester could improve maternal healthcare and in the long run reduce adverse outcomes for Swedish women. A national first trimester pregnancy biobank would facilitate future research on prevention and prediction of pregnancy complications.

A total of 13000 enrolled individuals will be needed for creating the model and for validation.

ELIGIBILITY:
Inclusion Criteria:

* Women with a Swedish personal identity number, who adhere to maternal care program before the end of the first trimester and have a planned first trimester scan (weeks 11-13) are eligible for the study.

Exclusion Criteria:

* Maternal age <18 years or language-barrier despite interpreter and written information.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — pregnant women
Study Population: All women attending a first trimester ultrasound at the study sites, which involves both tertiary as well as secondary hospitals and out-patient clinics.
Sampling Method: Non-Probability Sample
Enrollment: 13000 (Actual)
Dates: Start 2018-11-09 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Preterm Preeclampsia | delivery <37 gestational weeks
  Preeclampsia according to the Swedish definition, currently new onset hypertension (blood pressure ≥ 140/90) and proteinuria after gestational week 20.

SECONDARY OUTCOMES:
Small for gestational age | at delivery
  birthweight ≤ - 2 SD according to the Swedish reference curve
Overall preeclampsia | At delivery
  Preeclampsia according to the Swedish definition, currently new onset hypertension (blood pressure ≥ 140/90) and proteinuria after gestational week 20.
Preterm preeclampsia | delivery <37 gestational weeks
  Preeclampsia according to the Swedish definition prior to 2020 as well as the definition hereafter
Term preeclampsia | delivery >/=37 gestational weeks
  Preeclampsia according to the Swedish definition prior to 2020 as well as the definition hereafter

CONTACTS AND LOCATIONS:
Overall Officials: Lina Bergman, MD, PhD, Study Chair — Uppsala University; Peter Lindgren, MD, PhD, Study Chair — Karolinska Institutet; Anna Sandström, MD, PhD, Study Chair — Karolinska Institutet; Peter Conner, Ass Prof, Study Chair — Karolinska Institutet; Marius Kublickas, Ass Prof, Study Chair — Karolinska Institutet; Stefan Hansson, Professor, Study Chair — Lund University
Locations (9):
- Sweden (9):
  - Eskilstuna hospital, Eskilstuna, Sörmland
  - Södra Älvsborgs sjukhus, Borås, Västra Götalandsregionen
  - Norra Älvsborgs sjukhus, Trollhättan, Västra Götalandsregionen
  - County Council Dalarna, Falun
  - Gothenburg University, Sahlgrenska academy, dept of obstetrics and gynecology, Gothenburg
  - Lund University Hospital, dept of obstetrics and gynecology, Lund
  - Örebro University Hospital, Örebro
  - Karolinska Institute, Stockholm
  - Uppsala University Hopsital, department of women's and children's health, Uppsala

IPD SHARING:
Plan to Share IPD: Yes
There is a plan to make IPD and related data dictionaries available with a similar project in Denmark.
Supporting Information: CSR
Time Frame: 2021
Access Criteria: The steering committee will review requests. Requests can be sent to:
  Anna-karin.wikstrom@kbh.uu.se or ylva.carlsson@vgregion.se
URL: http://www.impactstudien.se

REFERENCES:
- [Result] Duley L. The global impact of pre-eclampsia and eclampsia. Semin Perinatol. 2009 Jun;33(3):130-7. doi: 10.1053/j.semperi.2009.02.010. PMID 19464502
- [Result] Mol BWJ, Roberts CT, Thangaratinam S, Magee LA, de Groot CJM, Hofmeyr GJ. Pre-eclampsia. Lancet. 2016 Mar 5;387(10022):999-1011. doi: 10.1016/S0140-6736(15)00070-7. Epub 2015 Sep 2. PMID 26342729
- [Result] Wikstrom AK, Larsson A, Eriksson UJ, Nash P, Norden-Lindeberg S, Olovsson M. Placental growth factor and soluble FMS-like tyrosine kinase-1 in early-onset and late-onset preeclampsia. Obstet Gynecol. 2007 Jun;109(6):1368-74. doi: 10.1097/01.AOG.0000264552.85436.a1. PMID 17540809
- [Result] Wright D, Syngelaki A, Akolekar R, Poon LC, Nicolaides KH. Competing risks model in screening for preeclampsia by maternal characteristics and medical history. Am J Obstet Gynecol. 2015 Jul;213(1):62.e1-62.e10. doi: 10.1016/j.ajog.2015.02.018. Epub 2015 Feb 25. PMID 25724400
- [Result] Akolekar R, Syngelaki A, Poon L, Wright D, Nicolaides KH. Competing risks model in early screening for preeclampsia by biophysical and biochemical markers. Fetal Diagn Ther. 2013;33(1):8-15. doi: 10.1159/000341264. Epub 2012 Aug 16. PMID 22906914
- [Result] Rolnik DL, Wright D, Poon LC, O'Gorman N, Syngelaki A, de Paco Matallana C, Akolekar R, Cicero S, Janga D, Singh M, Molina FS, Persico N, Jani JC, Plasencia W, Papaioannou G, Tenenbaum-Gavish K, Meiri H, Gizurarson S, Maclagan K, Nicolaides KH. Aspirin versus Placebo in Pregnancies at High Risk for Preterm Preeclampsia. N Engl J Med. 2017 Aug 17;377(7):613-622. doi: 10.1056/NEJMoa1704559. Epub 2017 Jun 28. PMID 28657417
- [Result] Mosimann B, Pfiffner C, Amylidi-Mohr S, Risch L, Surbek D, Raio L. First trimester combined screening for preeclampsia and small for gestational age - a single centre experience and validation of the FMF screening algorithm. Swiss Med Wkly. 2017 Aug 25;147:w14498. doi: 10.4414/smw.2017.14498. eCollection 2017. PMID 28871576
- [Result] Oliveira N, Magder LS, Blitzer MG, Baschat AA. First-trimester prediction of pre-eclampsia: external validity of algorithms in a prospectively enrolled cohort. Ultrasound Obstet Gynecol. 2014 Sep;44(3):279-85. doi: 10.1002/uog.13435. Epub 2014 Aug 13. PMID 24913190
- [Result] O'Gorman N, Wright D, Syngelaki A, Akolekar R, Wright A, Poon LC, Nicolaides KH. Competing risks model in screening for preeclampsia by maternal factors and biomarkers at 11-13 weeks gestation. Am J Obstet Gynecol. 2016 Jan;214(1):103.e1-103.e12. doi: 10.1016/j.ajog.2015.08.034. Epub 2015 Aug 19. PMID 26297382
- [Result] WHO Recommendations for Prevention and Treatment of Pre-Eclampsia and Eclampsia. Geneva: World Health Organization; 2011. Available from http://www.ncbi.nlm.nih.gov/books/NBK140561/ PMID 23741776
- [Result] Lindqvist PG, Molin J. Does antenatal identification of small-for-gestational age fetuses significantly improve their outcome? Ultrasound Obstet Gynecol. 2005 Mar;25(3):258-64. doi: 10.1002/uog.1806. PMID 15717289
- [Result] Sreeja Sarojini AG, Andrew Pecora and K. Stephen Suh. Proactive Biobanking to Improve Research and Health Care. Journal of Tissue Science & Engineering.
- [Result] Stephansson O, Petersson K, Bjork C, Conner P, Wikstrom AK. The Swedish Pregnancy Register - for quality of care improvement and research. Acta Obstet Gynecol Scand. 2018 Apr;97(4):466-476. doi: 10.1111/aogs.13266. Epub 2017 Dec 14. PMID 29172245
- [Derived] Bergman L, Sandstrom A, Jacobsson B, Hansson S, Lindgren P, Larsson A, Imberg H, Conner P, Kublickas M, Carlsson Y, Wikstrom AK. Study for Improving Maternal Pregnancy And Child ouTcomes (IMPACT): a study protocol for a Swedish prospective multicentre cohort study. BMJ Open. 2020 Sep 23;10(9):e033851. doi: 10.1136/bmjopen-2019-033851. PMID 32967865